CLINICAL TRIAL: NCT02292251
Title: Study to Enhance Motor Acute Recovery With Intensive Training After Stroke
Acronym: SMARTS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Columbia University (Other); University of Zurich (Other); James S McDonnell Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00047647
Record Dates: First submitted 2014-11-08; First posted 2014-11-17 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: Stroke; Transcranial direct current stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device-assisted therapy (Active Comparator): 30 hours of therapy with the ArmeoPower device, a commercially available device for arm rehabilitation
  Interventions: Behavioral: Device-assisted therapy
- Therapy-based occupational therapy (Active Comparator): 30 hours of conventional occupational therapy that emphasizes task-oriented training.
  Interventions: Behavioral: Therapy-based occupational therapy

INTERVENTIONS:
Behavioral: Device-assisted therapy
  Arms: Device-assisted therapy
Behavioral: Therapy-based occupational therapy
  Arms: Therapy-based occupational therapy

SUMMARY:
Stroke often results in limitation of arm movements, from which many people do not fully recover. We believe that early and intensive therapy is important to enhance recovery of arm movements after stroke. We are doing this research study to see how much arm movements improve with intensive therapy in patients have had a stroke in the past 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 21 years
2. Ischemic stroke confirmed by CT or MRI within the previous 6 weeks
3. No history of prior ischemic or hemorrhagic stroke with associated motor deficits (prior stroke with no motor symptoms is allowed)
4. Residual unilateral arm weakness with Fugl-Meyer Upper Extremity (FM-UE) score 6-40 at time of enrollment.
5. Ability to give informed consent and understand the tasks involved.

Exclusion Criteria:

1. Space-occupying hemorrhagic transformation or associated intracranial hemorrhage.
2. Arm impairment that is too severe or too mild on day of baseline testing just prior to beginning of the study intervention.
3. Recent botox injection to upper limb or planned botox injection over the course of the 7-month study duration.
4. Cognitive impairment, with score on Montreal Cognitive Assessment (MoCA) ≤ 20.
5. History of physical or neurological condition that interferes with study procedures or assessment of motor function (e.g. severe arthritis, severe neuropathy, Parkinson's disease).
6. Inability to sit in a chair and perform upper limb exercises for one hour at a time.
7. Participation in another upper extremity rehabilitative therapy study during the study period.
8. Terminal illness
9. Social and/or personal circumstances that interfere with ability to return for therapy sessions and follow up assessments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity (FM-UE) | from baseline to day 3 post-training
  Change in arm impairment, measured by FM-UE

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity (FM-UE) | from baseline to day 90 post-training
  Change in arm impairment, measured by FM-UE

CONTACTS AND LOCATIONS:
Overall Officials: John W. Krakauer, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University, New York, New York
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Krakauer JW, Kitago T, Goldsmith J, Ahmad O, Roy P, Stein J, Bishop L, Casey K, Valladares B, Harran MD, Cortes JC, Forrence A, Xu J, DeLuzio S, Held JP, Schwarz A, Steiner L, Widmer M, Jordan K, Ludwig D, Moore M, Barbera M, Vora I, Stockley R, Celnik P, Zeiler S, Branscheidt M, Kwakkel G, Luft AR. Comparing a Novel Neuroanimation Experience to Conventional Therapy for High-Dose Intensive Upper-Limb Training in Subacute Stroke: The SMARTS2 Randomized Trial. Neurorehabil Neural Repair. 2021 May;35(5):393-405. doi: 10.1177/15459683211000730. Epub 2021 Mar 20. PMID 33745372
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411